CLINICAL TRIAL: NCT07238959
Title: Application of Quantum Detection-Driven Artificial Intelligence Algorithms for Single-Molecule cfDNA Characterization in the Early Diagnosis of Prostate Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: West China Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); First Affiliated Hospital of Ningbo University (Network); Jiangsu Provincial People's Hospital (Other); The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Ren Shancheng, Professor, Chief of Urology, Shanghai Changzheng Hospital
Other Study IDs: CAPS
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Benign Prostate Hypertrophy(BPH); Prostate Cancer (Diagnosis); Prostate Neoplasm
Keywords: Early diagnosis; cfDNA
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study will extract and analyze cell-free DNA (cfDNA) from participants' peripheral blood. The study protocol does not plan for the long-term retention of any biospecimens. Upon completion of the cfDNA analysis, all remaining DNA samples will be securely disposed of. Only the de-identified derived data from the analyses will be retained for statistical analysis in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retrospective Testing Cohort
  Interventions: Diagnostic Test: Quantum Detection
- Prospective Internal Validation Cohort
  Interventions: Diagnostic Test: Quantum Detection
- Prospective external Validation Cohort
  Interventions: Diagnostic Test: Quantum Detection

INTERVENTIONS:
Diagnostic Test: Quantum Detection — This cohort will utilize archived plasma samples from a historical patient population with confirmed diagnoses (prostate cancer vs. controls). The objective is model development. The intervention involves analyzing these stored samples using the quantum sensing platform to extract multi-modal cfDNA features (e.g., fragmentomics, methylation). This data is then used to train and optimize the initial AI diagnostic algorithm, establishing the core model before prospective validation.
  Groups: Retrospective Testing Cohort
Diagnostic Test: Quantum Detection — This cohort will prospectively enroll new patients with suspected prostate cancer from the same institution as testing cohort. The objective is initial model validation. The intervention entails collecting pre-biopsy blood samples from these participants. The cfDNA from these fresh samples is analyzed using the locked model from the training phase. The model's predictions are then compared against the gold-standard prostate biopsy results to assess initial diagnostic performance.
  Groups: Prospective Internal Validation Cohort
Diagnostic Test: Quantum Detection — This cohort will prospectively recruit patients from multiple independent clinical centers. The objective is to test the model's generalizability. The intervention involves standardized blood collection across all external sites, with samples sent to a central lab for blinded cfDNA analysis using the finalized, locked-down model.
  Groups: Prospective external Validation Cohort

SUMMARY:
This research project aims to develop a novel blood testing method integrating cutting-edge quantum sensing and artificial intelligence technologies to achieve precise, non-invasive early diagnosis of prostate cancer. The research will employ quantum sensors to perform ultra-high-sensitivity measurements of circulating free DNA (cfDNA) in blood, thereby training a dedicated AI diagnostic model. The ultimate objective is to establish the diagnostic efficacy of this approach through clinical validation, providing clinicians with a novel diagnostic tool capable of significantly reducing unnecessary prostate biopsy procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Male, aged 18-80 years;
2. PSA > 4 ng/ml;
3. Patients meeting criteria for prostate biopsy:

   * fPSA/PSA < 0.16 or PSA D > 0.15 or PSA V > 0.75; ② Positive digital rectal examination (DRE); ③ Imaging studies (ultrasound/MRI) showing suspicious lesions.

Exclusion Criteria:

1. Patients diagnosed with any malignant tumour within the past five years;
2. Patients who have undergone transurethral resection or enucleation of the prostate;
3. Patients who have previously received treatment for prostate cancer, including but not limited to endocrine therapy, targeted therapy, or immunotherapy;
4. Patients on long-term anticoagulant or antiplatelet therapy (anticoagulants discontinued for less than one week);
5. Patients who have received any form of tumour treatment prior to enrolment blood sampling, including surgery, radiotherapy/chemotherapy, endocrine therapy, targeted therapy, or immunotherapy;
6. Concurrent severe systemic diseases deemed by the investigator likely to interfere with trial treatment, evaluation, or compliance, including serious respiratory, circulatory, neurological, psychiatric, gastrointestinal, endocrine, immunological, or urological disorders;
7. Organ transplant recipients or individuals with prior non-autologous (allogeneic) bone marrow or stem cell transplantation;
8. Subjects who have undergone blood transfusion within one month prior to blood sampling;
9. Patients currently participating in other clinical trials, or who have participated in other clinical trials within the past year;
10. Patients deemed unsuitable for this clinical trial by the investigator;
11. Patients meeting any of the above criteria shall not be eligible for inclusion as subjects.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males aged 18-80 years with elevated PSA (>4 ng/ml) and clinical indications for prostate biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve (AUC-ROC) for the predictive model in the general population for prostate cancer. | Through primary completion which may take 12 months.
Sensitivity of the predictive model in detecting prostate cancer within the general population. | Through primary completion which may take 12 months.
Specificity of the predictive model in detecting prostate cancer within the general population. | Through primary completion which may take 12 months.

SECONDARY OUTCOMES:
Area under the ROC curve for the predictive model in identifying prostate cancer within the PSA grey zone cohort. | Through primary completion which may take 12 months.
Sensitivity of the predictive model in identifying prostate cancer within the PSA grey zone cohort. | Through primary completion which may take 12 months.
The specificity of the predictive model in identifying prostate cancer among individuals in the PSA grey zone. | Through primary completion which may take 12 months.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Aﬃliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Ningbo No. 1 Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No